CLINICAL TRIAL: NCT05503056
Title: The Utilization of Art Therapy During Pregnancy to Reduce the Incidence of Postpartum Depression
Brief Title: Art Therapy in Obstetric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Sara N. Iqbal, Primary Investigator, Medstar Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20223247
Record Dates: First submitted 2022-03-20; First posted 2022-08-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related; Depression
MeSH Terms: conditions — Depression | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Engage in six art therapy sessions
  Interventions: Other: art therapy
- Control (Placebo Comparator): Engage in usual activities
  Interventions: Other: nothing

INTERVENTIONS:
Other: art therapy — six sessions of art therapy with licensed therapists
  Arms: Intervention
Other: nothing — no intervention to this group
  Arms: Control

SUMMARY:
This is a prospective study examining the potential impact art therapy has on postpartum depression and mother-baby bonding in women. Women who receive care at Washington Hospital Center's will be recruited for this study.

DETAILED DESCRIPTION:
The purpose of this research study is to assess whether alternative mental health interventions positively impacts maternal-infant bonding and postpartum depression rates in women. Postpartum depression continues to be a prevalent concern for mothers and families in the United States, with current estimates demonstrating 10-20% of women being diagnosed within one year of birth. The risks of developing postpartum depression are not well known, with maternal anxiety and stress during pregnancy being one of the proposed predisposing factors. Women with high-risk pregnancies are particularly susceptible to higher levels of stress and depression, during their pregnancy thus leaving them at great risk for postnatal depression. Given this association, finding ways to alleviate stressors is important.

Music therapy is a known intervention linked with improved outcomes in women undergoing procedural interventions, including labor and delivery. Art therapy is also associated with improved outcomes, though outside of obstetrics. In elderly women with depression and those with breast cancer diagnoses, visual art therapy has been shown to be superior to other non-medicinal interventions in improving mood. Current data is both qualitative as well as quantitative, demonstrating positive impacts on patients.

While evidence exists to support the utilization of these alternative forms of therapy, they have not been adequately applied to pregnant and postpartum women outside of music therapy. With the understanding that other art forms are tied with improvement in anxiety, depression, and quality of life, the implementation in this special patient population is paramount. Investigating how a relatively benign intervention can possibly promote improvement in maternal mental health, thus allowing for better mother-baby bonding in the first year of life, is key in finding ways to support the growth and development of healthy families.

ELIGIBILITY:
Inclusion Criteria:

* Participants will have to be eighteen years of age or older
* in the second trimester of pregnancy at time of recruitment
* speak and read English as their primary language
* have access to a reliable internet/wifi connection to participate in therapy sessions
* plan to deliver at Washington Hospital Center

Exclusion Criteria:

- Women who do not meet those criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-04-13 (Actual)

PRIMARY OUTCOMES:
changes in Edinburgh Postnatal Depression Scale scores | start, and end of intervention period; time of delivery, two weeks postpartum, six weeks postpartum, three months postpartum
  raw score on scale
change in maternal-infant bonding scores | start, and end of intervention period; time of delivery, two weeks postpartum, six weeks postpartum, three months postpartum
  raw score on scale
utilization of behavioral health/psychology/psychiatry services during pregnancy and postpartum | start, and end of intervention period; time of delivery, two weeks postpartum, six weeks postpartum, three months postpartum
  chart review to see if patients utilized services "yes" vs. "no"
use of psychiatry medications during and after pregnancy | start, and end of intervention period; time of delivery, two weeks postpartum, six weeks postpartum, three months postpartum
  chart review to see if patients utilized services "yes" vs. "no"

SECONDARY OUTCOMES:
obstetrical complications (postpartum hemorrhage, OASIS, ICU admission) | up to 3 months postpartum
  chart review
gestational age at time of delivery | delivery
  chart review
mode of delivery | delivery
  chart review
reason for delivery (iatrogenic vs spontaneous) | delivery
  chart review
birth weight | delivery
  chart review
APGAR scores | delivery
  chart review
NICU admissions | delivery
  chart review
delivery complications (shoulder dystocia, low birth weight) | delivery
  chart review

CONTACTS AND LOCATIONS:
Overall Officials: Sara N Iqbal, MD, Principal Investigator — MedStar Health
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciasca EC, Ferreira RC, Santana CLA, Forlenza OV, Dos Santos GD, Brum PS, Nunes PV. Art therapy as an adjuvant treatment for depression in elderly women: a randomized controlled trial. Braz J Psychiatry. 2018 Jul-Sep;40(3):256-263. doi: 10.1590/1516-4446-2017-2250. Epub 2018 Feb 1. PMID 29412335